CLINICAL TRIAL: NCT05042219
Title: The Relationship Between Pulmonary and Cardiac Dysfunction and the Cardiac Effects of Pulmonary Treatments: Cardiopulmonary MRI Analysis
Brief Title: Effects of Pulmonary Diseases and Their Treatment on Cardiac Function
Status: Recruiting | Type: Observational
Sponsor: Ayham Daher (Other)
Responsible Party: Sponsor-Investigator, Ayham Daher, Principal Investigator, RWTH Aachen University
Organization: RWTH Aachen University (Other)
Other Study IDs: Uniklinik RWTH Aachen
Record Dates: First submitted 2021-09-02; First posted 2021-09-13 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: COPD; Bronchial Asthma; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Idiopathic Pulmonary Fibrosis | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- COPD (ICS): COPD before initiation of inhaled corticosteroid therapy
  Interventions: Diagnostic Test: Cardiac MRI
- COPD (LTOT-NIV): COPD before initiation of long term oxygen therapy or domiciliary long-term non-invasive ventilation
  Interventions: Diagnostic Test: Cardiac MRI
- COPD (Roflumilast ): COPD before initiation of Roflumilast therapy
  Interventions: Diagnostic Test: Cardiac MRI
- Bronchial asthma (antibody): Bronchial asthma before initiation of antibody therapy
  Interventions: Diagnostic Test: Cardiac MRI
- Bronchial asthma (ICS): Bronchial asthma before initiation of inhaled corticosteroid therapy
  Interventions: Diagnostic Test: Cardiac MRI
- Pulmonary fibrosis: Pulmonary fibrosis before initiation of antifibrotic therapy
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Cardiac MRI and Echocardiography before treatment initiation of pulmonary disease and 3 months thereafter
  Other Names: Echocardiography

SUMMARY:
While the bidirectional relationship between the lung and the right heart are well studied, the cardiopulmonary interactions between the lung and the left heart are largely unresearched and not well understood. However, in recent years, there is a growing evidence that partially explains the bidirectional interaction between COPD and left heart. Systemic inflammation with multiorgan involvement is thought to play a role in COPD as a systemic disease. Some therapeutic approaches to COPD also appear to influence these cardiopulmonary interactions. While understanding these interactions is very important for clinicians, scientific data are scarce. Cardiac magnetic resonance imaging (cardiac MRI) is the gold standard for assessing cardiac function and dimensions as well as myocardial inflammation. Despite this excellent suitability of cardiac MRI for the assessment of cardiovascular function, only few studies have investigated cardiac function and myocardial structure in patients with pulmonary disease using cardiac MRI. Such a study is therefore very important for understanding the effects of pulmonary disease and its management on the heart.

The objective is to determine cardiac function in patients with pulmonary disease and to analyze the cardiovascular effects of the treatment of the pulmonary disease.

Specifically, the following will be studied:

* Using cardiac MRI: Cardiac function and volumes and indications of myocardial fibrosis and edema in patients with chronic pulmonary disease at the time of first diagnosis.
* the vascular function of pulmonary arteries in these patients, also using cardiac MRI
* the relationship between pulmonary function parameters and cardiac dysfunction to identify patients at increased risk, if applicable.
* Echocardiographic assessment of left heart including strain analysis.
* the course of these cardiovascular parameters (using cardiac MRI and echocardiography) 3-6 months after initiation of guideline-based therapy for pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic lung disease requiring treatment (COPD, asthma, or pulmonary fibrosis).
* Age > 18 years
* Informed consent to participate in the study will sign

Exclusion Criteria:

* Individuals who are not fully capable of giving consent and understanding the nature, significance and scope of the study.
* Patients with contraindications to MRI examination (eg, pacemaker, severe claustrophobia) or to contrast medium use (severe renal insufficiency or glomerular filtration rate <30 ml/min, known gadolinium contrast medium allergy)
* Patients with atrial fibrillation or other significant cardiac arrhythmias that interfere with cardiac MRI
* Pregnancy and lactation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with COPD group D and new prescription of ICS therapy.
  * Patients with COPD and new prescription of long-term O2 therapy or domiciliary long-term non-invasive ventilation.
  * Patients with COPD and new prescription of Roflumilast therapy.
  * Patients with bronchial asthma and new prescription of antibody therapy.
  * Patients with bronchial asthma at initial diagnosis and new prescription of ICS mono-therapy.
  * Patients with initial diagnosis of pulmonary fibrosis and new prescription of antifibrotic therapy (nintedanib or pirfinidone).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-09-14 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
left-ventricular end-diastolic volume | 3 months
  left-ventricular end-diastolic volume before and after therapy

SECONDARY OUTCOMES:
Pulmonary microvascular blood flow (physiological parameter: ml/min/100 ml Lung volume) | 3 months
  Pulmonary microvascular blood flow (physiological parameter: ml/min/100 ml Lung volume) before and after therapy
Presence of myocardial fibrosis or edema (pathophysiological parameter: yes/no) | 3 months
  Presence of myocardial fibrosis or edema (pathophysiological parameter: yes/no) before and after therapy
Left ventricular global longitudinal strain (physiological parameter) | 3 months
  Left ventricular global longitudinal strain (physiological parameter) before and after therapy

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Undecided